CLINICAL TRIAL: NCT03309111
Title: A Phase 1, First-in-Human, Multicenter, Open-Label, Two-Part Dose-Escalation and Cohort Expansion Study of Single-Agent ISB 1342 in Subjects With Previously Treated Multiple Myeloma
Brief Title: Study of ISB 1342, a CD38/CD3 Bispecific Antibody, in Subjects With Previously Treated Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ichnos Sciences SA (Industry)
Collaborators: Glenmark Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISB 1342-101; 2016-005253-20 (EudraCT Number)
Record Dates: First submitted 2017-10-04; First posted 2017-10-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ISB 1342 (Experimental): Part 1: Cohorts of multiple ISB 1342 dose levels; Part 2: One dose regimen until disease progression or other discontinuation criterion is met
  Interventions: Biological: ISB 1342

INTERVENTIONS:
Biological: ISB 1342 — ISB-1342 is CD38 x CD3 BEAT® 1.0 bispecific antibody. ISB 1342 is administered by intravenous (IV) infusion or subcutaneous injection (SC)

SUMMARY:
The purpose of this study is to assess safety, efficacy, pharmacokinetic (PK)/pharmacodynamic (PD), and immunogenicity with ISB 1342 in subjects with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
This study is an open-label, multi-center, Phase 1 study of ISB 1342 in subjects with relapsed/refractory multiple myeloma refractory to proteasome inhibitors (PIs), immunomodulators (IMiDs), and daratumumab. There will be a dose escalation phase (Part 1) and dose expansion phase (Part 2). In Part 1 of the study, subjects will be treated at escalating dose levels. Once the recommended part 2 dose (RP2D) of ISB 1342 is declared in Part 1, the expansion phase (Part 2) will be initiated at the RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of multiple myeloma with measurable disease (serum, urine, or free light chain) per International Myeloma Working Group (IMWG) criteria, including non-secretory or oligo-secretory multiple myeloma which has relapsed after or is refractory to prior therapies, including proteasome inhibitors (PIs), immunomodulators (IMiDs) and anti-CD38 targeted therapies (daratumumab, isatuximab).
* Eastern Cooperative Oncology Group (ECOG) performance-status score of 2 or less and 1 or less (for France).
* Adequate hematologic, renal, and hepatic functions
* Seronegative for hepatitis B antigen; positive hepatitis B tests can be further evaluated by confirmatory tests, and if viral load is negative, the subject can be enrolled.
* Seronegative for hepatitis C antibody; if positive, then further test for the presence of antigen by hepatitis C virus polymerase chain reaction (HCV PCR). If HCV antigen tests are negative, then the subject can be enrolled.
* Oxygen saturation level ≥92% on room air.
* Left ventricular ejection fraction (LVEF) ≥50% and no pericardial or pleural effusion at Screening

Exclusion Criteria:

* Active central nervous system involvement
* Exposure to daratumumab or isatuximab within 2 months prior to the start of study treatment
* Active plasma cell leukemia
* Active infectious disease
* Clinically significant cardiovascular and respiratory conditions
* History of HIV infection
* Subjects requiring prohibited concomitant medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated dose (MTD) and/or recommended part 2 dose (RP2D) of ISB 1342 (Part 1) | 28 days
Proportion of subjects with an investigator-assessed objective response (at least a partial response or better), complete response, disease control (stable disease or better) to ISB 1342, per International Myeloma Working Group (IMWG) criteria (Part 2) | 28 days

SECONDARY OUTCOMES:
Number of subjects with adverse events based on frequency and severity as assessed by common terminology criteria for adverse events (CTCAE) v5.0 (Part 1 and Part 2) | up to 30 days post last dose
Maximum serum concentration (Cmax) of ISB 1342 (Part 1 and Part 2) | 28 days
Time to reach maximum observed plasma concentration (Tmax) of ISB 1342 (Part 1 and Part 2) | 28 days
Area under the serum concentration time curve from zero to time t (AUC0-t) of ISB 1342 (Part 1 and Part 2) | 28 days
Area under the curve from time zero to end of dosing interval (AUC0-tau) of ISB 1342 (Part 1 and Part 2) | 28 days
Immunogenicity of ISB 1342 by anti-drug antibody (ADA) formation (Part 1 and Part 2) | 28 days
Percent incidence of neutralizing antibody formation from positive anti-drug antibody (ADA) samples assessed from baseline until end of treatment (EOT) (Part 1 and Part 2) | 28 days
Efficacy of ISB 1342 (duration of response [DOR]) (Part 1 and Part 2) | 28 days
Efficacy of ISB 1342 (disease control rate [DCR]) (Part 1 and Part 2) | 28 days
Efficacy of ISB 1342 (duration of disease control) (Part 1 and Part 2) | 28 days
Efficacy of ISB 1342 (time to minimal residual disease [MRD] negative status) (Part 1 and Part 2) | 28 days
Efficacy of ISB 1342 (progression free survival [PFS]) (Part 2) | 28 days
Efficacy of ISB 1342 (time to treatment failure [TTF]) (Part 2) | 28 days
Efficacy of ISB 1342 (time to disease progression [TTP]) (Part 2) | 28 days
Efficacy of ISB 1342 (overall survival [OS]) (Part 2) | Time from first dose until death from any cause or end of study collection, whichever is later, assessed up to 60 months.
Proportion of subjects with investigator-assessed objective response (at least a partial response or better), complete response, disease control (stable disease or better) to ISB 1342, per International Myeloma Working Group (IMWG) criteria (Part 1) | 28 days

CONTACTS AND LOCATIONS:
Locations (20):
- United States (9):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Johns Hopkins Medicine - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Mayo Clinic Cancer Center (MCCC) - Rochester, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai Beth Israel, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke Clinical Research Institute, Durham, North Carolina
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
- France (11):
  - CHU de Nantes - Hôtel-Dieu, Nantes, Cedex
  - CHU Hopitaux de Bordeaux - Hôpital Haut-Lévêque, Pessac, Cedex
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite, Cedex
  - CHU de Poitiers, Poitiers, Cedex
  - CHU de Rennes - Hôpital Pontchaillou, Rennes, Cedex
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse, Cedex
  - CHRU de Tours - Hôpital Bretonneau, Tours, Cedex
  - CHU Hôpital Henri Mondor, Créteil
  - Centre Hospitalier Régional Universitaire de Lille (CHRU) - Hôpital Claude Huriez, Lille
  - L'Institut Paoli - Calmettes, Marseille
  - Hôpital Saint-Antoine, Paris

IPD SHARING:
Plan to Share IPD: No